CLINICAL TRIAL: NCT05010720
Title: Prevelance of Frailty and Its Associated Factors in Patients With Axial Spondyloarthritis
Status: Completed | Type: Observational
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Özgül Öztürk, Assistant Professor, Acibadem University
Other Study IDs: ATADEK 2021/14
Record Dates: First submitted 2021-08-12; First posted 2021-08-18 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Frailty; Axial Spondyloarthritis
MeSH Terms: conditions — Frailty; Axial Spondyloarthritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Axial Spondyloarthritis is an inflammatory arthritis disease and its main symptoms are chronic pain and stiffness, causing structural damage to the spinal vertebrae. Axial Spondyloarthritis leads to physical disability and a decrease in the level of physical activity.

Frailty is a syndrome characterized by decline in physiological reserve and loss of muscle strength. Frailty can lead to vulnerability of individuals to possible injuries and a decrease in independence, and ultimately an increase in mortality. Although frailty is associated with older adults, it has been reported that it can be detected in patients with cancer, diabetes and rheumatological diseases and it is not related with age. Frailty has been reported to be a reversible and a treatable condition.

The aim of our study was to investigate the prevalence of frailty and the relationship between frailty and disease activity, physical functional level, quality of life and other associated factors in individuals with Axial Spondyloarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Axial Spondyloarthritis by an experienced rheumatologist.
* To be between the ages of 40-65

Exclusion Criteria:

* Severe comorbidities such as cancer and stroke
* Being diagnosed with newly defined or recurrent cancer,
* Not having enough cognitive skills to answer the questions,
* Having neurological problems such as stroke
* Having cognitive impariment

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Axial Spondyloarthritis in a tertiary research and training hospital
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-08-12 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Fried Frailty Phenotype | 1 day
  The frailty level of the participants included in the study will be determined according to the frailty phenotype criteria of Fried et al. criteria for the diagnosis of frailty; Decreased grip strength, walking speed for 4 meters is less than the determined metrics ( for people who are 159 cm and shorter as <6.12 sec or >5.25 sec for those 159 cm and above), involuntary weight loss in the last year (≥4.5 kg) or body mass index ≤18.5 kg/m2, low physical activity level, and increased fatigue level reported by the participant. Individuals meeting 3 or more of these criteria are defined as "frail", individuals meeting 1 or 2 criteria are defined as "pre-fragile (pre-fragile) and individuals who do not meet any criteria are defined as "normal or robust".
Kihon Checklist | 1 day
  Frailty status will determined according to the Turkish version of the Kihon Checklist (KCL) which consists of 25 questions for yes (1) or no (0) answers. KCL includes seven categories as; physical function (5 items), mood (5 items), instrumental activities of daily life (5 items), nutrition (2 items), oral function (3 items), memory (3 items) and socialization (2 items). Total KCL scores range from 0 to 25 and scores ≥8 indicate frailty, between 4 to 7 indicate pre-frailty and between 0 to 3 indicate robustness.
Short Physical Performance Battery(SPPB) | 1 day
  SPPB can be used to determine frailty status. It comprises 3 parameters: static balance, sit to stand test and walking speed. Scores above 9 indicates no frailty, between 7 to 9 indicates pre-frailty and below 7 indicates frailty status.

SECONDARY OUTCOMES:
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | 1 day
  BASDAI evaluates disease-specific symptoms such as fatigue, joint pain, and morning stiffness in individuals with Ankylosing Spondylitis between 0 and 10. A high score is expressed by an increase in disease activity.
Bath Ankylosing Spondylitis Functional Index (BASFI) | 1 day
  BASFI has been developed to determine the functional status of individuals with Ankylosing Spondylitis and evaluates the perceived stress level in daily activities between 0 and 10 (0 = easy and 10 = impossible). Activities such as bending, reaching, standing, changing positions, climbing stairs are questioned. The total score is determined by dividing the sum of the scores from each item by 10, and "0" is defined as the best score and "10" as the worst score.
Depression and Anxiety | 1 day
  Depression and anxiety status of the included patients will be evaluated with the Turkish version of the Hospital Anxiety and Depression Scale (HADS). This scale consists of 14 items; 7 for depression symptoms and 7 for anxiety symptoms. Each answer is scored 0 to 3. Cut-off values for the Turkish version are 7 and 10 for depression and anxiety subscales, respectively.
Ankylosing Spondylitis Quality of Life Scale | 1 day
  The Turkish version of the Ankylosing Spondylitis Quality of Life (ASQOL) scale will be used to assess disease-related quality of life. ASQOL includes 18 items with dichotomous responses (yes/no) evaluating the impact of disease on social life, sleep, motivation, mood, coping, independence and activities of daily living, The score ranges between 0 to 18 and higher score indicates reduced quality of life.

OTHER OUTCOMES:
Gait Speed | 1 day
  The patient will be asked to walk 4 meter distance in a normal gait speed for two times. The shortest time will be recorded.
Grip Strength | 1 day
  Grip strength will be evaluated with JAMAR dynamometer. The patient will be positioned in a chair with the elbow flexed to 90 degrees and the wrist in a neutral position, and he/she will be asked to grip as strong as he/she can do for 3 seconds. The test will be repeated 3 times and the highest value will be recorded.
Physical Activity Level | 1 day
  The physical activity level reported by the participants will be evaluated with the International Physical Activity Questionnaire - Short Form. The International Physical Activity Questionnaire - Short Form questions the time to spent in walking, moderate and vigorous activities, and sitting with 7 questions. The duration (minutes) and frequency (days) of each activity are questioned. According to the survey results, the physical activity levels of the participants will be classified as inactive, minimally active and very active.

CONTACTS AND LOCATIONS:
Locations (1):
- Haydarpaşa Numune Research and Training Hospital, Istanbul, Turkey (Türkiye)